CLINICAL TRIAL: NCT01700569
Title: Phase I Study of Escalated Pharmacologic Dose, of Oral Folinic Acid in Combination With Temozolomide, According to Stupp R. Regimen, in Patients With Operated Grade-IV Astocytoma and a Non-methylated Gene Status of MGMT.
Brief Title: Phase-1 Study of Folinic Acid to Modulate MGMT Gene in Glioblastoma
Acronym: FOLAGLI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: changing the standard of care
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Centre Antoine Lacassagne (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO 2012-02; 2012-000774-31 (EudraCT Number)
Record Dates: First submitted 2012-09-12; First posted 2012-10-04 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2021-05

CONDITIONS: Grade IV Astrocytoma; Glioblastoma
Keywords: high-grade; glioma; epigenetic
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Temozolomide; Particle Accelerators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Folinic Acid (Experimental): Folinic acid is given orally every day during the radiation therapy (47 days), then 5 days at each of the 6 maintenance cycle of temozolomide. The dose is escalated in a "3x3" method and the levels are: 5mg, 10mg, 15mg, 30mg, 60mg.
  Interventions: Drug: Temozolomide; Drug: folinic acid at pharmacological dose is the escalated drug; Radiation: High voltage radiation therapy (linear accelerator)

INTERVENTIONS:
Drug: Temozolomide — All the Patients are treated by oral Temozolomide 75 mg/m²/day every day during 42 days, 30 minutes after Folinic acid and 120 min before the radiation dose to the brain tumor. After one month rest, the maintenance phase consists of:Temozolomide is given orally (30 min after Folinic acid), at 200 mg/m²/day every day during 5 days: one course every month during 6 months (6 maintenance course).
  Other Names: Temodal; capsule dosage available: 5, 20, 10, 180 and 250 mg
Drug: folinic acid at pharmacological dose is the escalated drug
  Other Names: Folinate de Calcium, Lederfoline
Radiation: High voltage radiation therapy (linear accelerator) — Brain tumor field is irradiated Five days a week, during Stupp regimen during 6 weeks. During the sams time, Folinic acid and Temozolomide are given orally every days (six weeks).

SUMMARY:
O6-méthylguanine méthyltransférase (MGMT) is the main repair gene after DNA lesion induced by Temozolomide in combination with radiation therapy of Glioblastoma (GBM) in Stupp.R et al published regimen. In preclinical models, it has been demonstrated that MGMT methylation (which is silencing the DNA repair process) is achievable by folic acid. About half of the patients with operated GBM have an un-methylated MGMT gene status and therefore a poorer prognosis. A phase-1 dose escalation study is proposed with pharmacologic doses of folinic acid in combination with temozolomide and radiotherapy of operated GBM.

DETAILED DESCRIPTION:
Glioblastoma treated by Stupp regimen (Temozolomide + radiation therapy) have a different outcome depending on the methylation status of MGMT gene: when the gene is unmethylated, the repair process is active and the prognostic poor. In pre-clinical models, it has been demonstrated that Folic acid could re-methylate the MGMT gene and therefore the repair process to radiation and temozolomide could be limited, allowing a better prognosis. The proposed phase-1 study will explore the safety and efficacy of escalated doses of oral Folinic acid concomitantly with Stupp regimen. To determine the MTD is the main objective of the study, then the toxicty profile, the RDP2 and the methylation process efficacy at the MGMT gene level.

ELIGIBILITY:
Inclusion Criteria:

* Operated GBM (complete or near complete resection)
* Un-methylated MGMT gene

Exclusion Criteria:

* Non operable GBM
* Methylated MGMT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose | day 43
  maximal tolerated dose 3x3 patients inclusion(modified Fibonnacci dose escalation )

SECONDARY OUTCOMES:
MGMT gene re-methylation | day 43
  MGMT gene re-methylation in tumoral and blood samples

OTHER OUTCOMES:
Progression-free survival (PFS) | Year 1
  Progression-free survival (PFS)
Folic acid and Temozolomide combination Toxicity evaluation | day 43
  Acute toxicity: Common toxicity criteria version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Mario CAMPONE, MD, PhD, Principal Investigator — Institut Cancerologie de l'Ouest
Locations (4):
- France (4):
  - Institut de Cacerologie de l'ouest - site Paul Papin, Angers
  - CHU de Lyon, Bron
  - ICO site Gauducheau, Nantes
  - CLCC Antoine Lacassagne, Nice

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009